CLINICAL TRIAL: NCT07100496
Title: Evaluation of MIG-SPRAY Treatment on Migraine
Acronym: MIG-S
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RBHP 2024 PICKERING 2; 2024-A02815-42 (Other: ANSM)
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (MIG-SPRAY) (Experimental)
  Interventions: Combination Product: MIG-SPRAY
- Control group (no device) (No Intervention)

INTERVENTIONS:
Combination Product: MIG-SPRAY — MIG-SPRAY® is a film-forming liquid dressing designed for the preventive treatment of migraine.
  Key Features:
  * Administration:
    * Applied as 2 sprays per nostril, 3 times daily.
    * Treatment duration: 3 months.
  * Mechanism: Forms a protective film on the nasal mucosa, potentially modulating local triggers of migraine.
  * Use Case: Prophylactic (preventive) therapy for migraine, intended to reduce attack frequency and severity.
  Additional Notes:
  * Non-systemic (local action).
  * CE-marked as a Class I medical device (under EU Directive 93/42/EEC).
  Arms: Intervention group (MIG-SPRAY)

SUMMARY:
The goal of this clinical trial is to evaluate the real-world tolerability of the MIG-SPRAY device in adults aged 18-55 diagnosed with migraine (according to nternational Classification of Headache Disorders 3rd edition, code 1.1(ICHD-3)) for over 1 year.

The main questions it aims to answer are:

* Does MIG-SPRAY significantly reduce the composite score of expected adverse events (e.g., allergic reactions, nausea, headache) compared to no intervention, graded via a Likert scale (using the Common Terminology Criteria for Adverse Event (CTCAE v5.0))?
* Are there differences in unexpected adverse events, monthly migraine frequency, or Migraine Disability Assessment (MIDAS) scores between groups?

Researchers will compare the intervention group (MIG-SPRAY) to the control group (no device) to assess:

1. Tolerability (primary outcome).
2. Unexpected adverse events, migraine frequency, and disability (secondary outcomes).

Participants will:

* Be randomized (2:1) to MIG-SPRAY (n=30) or control (n=15).
* Use an electronic diary daily to report adverse events and migraine episodes.
* Complete the MIDAS questionnaire at baseline and post-treatment.
* Undergo monthly physician calls to review and grade adverse events.

Study design:

* Post-marketing, monocentric, open-label, randomized trial (Clermont-Ferrand University Hospital).
* Category 4.2 clinical investigation (CE-marked Class I device, used per labeling).
* No changes to background migraine therapy permitted.

Key eligibility:

* Age 18-55, migraine diagnosis ≥1 year (ICHD-3).
* Effective contraception (females of childbearing potential).
* Social security coverage and written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 55 years
* Migraine diagnosis for >1 year
* Meeting ICHD-3 (International Classification of Headache Disorders 3rd edition, code 1.1) diagnostic criteria
* Effective contraception for females of childbearing potential
* Sufficient cooperation and understanding to comply with trial requirements
* Provided informed consent after receiving complete study information
* Enrolled in the French Social Security system

Exclusion Criteria:

* Hypersensitivity: Known allergy to any component of the investigational product(s), salicylates, or camphor.
* Substance abuse: Current drug dependence or abuse (investigator's judgment).
* Pregnancy/breastfeeding: Pregnant or lactating women.
* Concurrent trials: Participation in another clinical trial, ongoing exclusion period, or receipt of >€6000 in trial-related compensation in the past 12 months.
* Legal protections: Under legal guardianship, curatorship, or deprivation of liberty.
* Medical incompatibility: Any condition deemed unsafe for participation (investigator's assessment).
* Significant medical history: Relevant comorbidities or antecedents (investigator's discretion).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The composite score of expected adverse events | From visit 1 (day 1) to the end of treatment (day 90)
  The study's primary endpoint is a composite score of adverse events (AEs) recorded during MIG-SPRAY® use.
  Key Details:
  - Calculation: Sum of severity grades (1-4 points, Likert scale) for 10 predefined AEs based on published device data: Allergic reaction, nausea, vomiting, dizziness, headache, drowsiness, sneezing, stomach pain, sore throat, and nasal dryness.
  * Grading: AEs are assessed via CTCAE v5.0 and aggregated into a single composite score.
  * Data Collection:
    * Patients report AEs daily via an electronic diary.
    * Study physicians monthly verify and grade AEs using the predefined Likert scale.
  Purpose: To quantitatively evaluate MIG-SPRAY®'s tolerability profile during the treatment period.

SECONDARY OUTCOMES:
Unexpected adverse events | From visit 1 (day 1) to the end of treatment (day 90)
  All adverse events (AEs) not previously listed as expected events, reported by patients in both the MIG-SPRAY® and control groups, will be recorded in a daily electronic diary.
  Key Assessment Criteria:
  * Any AE with a "possible" causal relationship to the study product (as determined by the investigator) will be classified as treatment-related
  * These unexpected AEs will be graded (1-4) using the NCI-CTCAE v5.0 Likert scale
  * A composite score will be calculated by summing the severity grades of all unexpected AEs during the treatment period
Number of migraine | From visit 1 (day 1) to the end of treatment (day 90)
  Patients will record all migraine episodes in a daily electronic diary throughout the treatment period. Data collection will cover the entire duration of product use.
Measurement of the Migraine Disability Assessment (MIDAS) | day 1
  The MIDAS questionnaire quantifies headache-related functional impairment through symptom intensity and quality-of-life impact metrics, categorizing patients into four distinct severity grades (I-IV) based on affected days. This patient-administered instrument facilitates evidence-based treatment stratification, with Grade I indicating minimal disability (0-5 days) and Grade IV representing significant impairment (>20 days).
Measurement of the Migraine Disability Assessment (MIDAS) | day 90
  The MIDAS questionnaire quantifies headache-related functional impairment through symptom intensity and quality-of-life impact metrics, categorizing patients into four distinct severity grades (I-IV) based on affected days. This patient-administered instrument facilitates evidence-based treatment stratification, with Grade I indicating minimal disability (0-5 days) and Grade IV representing significant impairment (>20 days).

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING,, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No